CLINICAL TRIAL: NCT00352300
Title: A Phase I Trial of Dose Dense (Biweekly) Carboplatin Combined With Paclitaxel and Pegfilgrastim (Neulasta): A Feasibility Study in Patients With Untreated Stage III and IV Ovarian, Tubal or Primary Peritoneal Cancer
Brief Title: Carboplatin, Paclitaxel, and Pegfilgrastim in Treating Patients With Stage III or Stage IV Ovarian Epithelial, Fallopian Tube, Primary Peritoneal, or Carcinosarcoma Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9919; NCI-2009-00622 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000486412; GOG-9919; GOG-9919 (Other: Gynecologic Oncology Group); GOG-9919 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Fallopian Tube Carcinoma; Infectious Disorder; Neutropenia; Ovarian Carcinosarcoma; Primary Peritoneal Carcinoma; Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Communicable Diseases; Neutropenia; Ovarian Neoplasms | interventions — Chemotherapy, Adjuvant; Carboplatin; Paclitaxel; Taxes; pegfilgrastim

ARMS (1):
- Treatment (carboplatin, paclitaxel, pegfilgrastim) (Experimental): Patients receive carboplatin IV and paclitaxel IV over 3 hours on day 1. Patients also receive pegfilgrastim subcutaneously on day 2.
  Interventions: Procedure: Adjuvant Therapy; Drug: Carboplatin; Drug: Paclitaxel; Biological: Pegfilgrastim

INTERVENTIONS:
Procedure: Adjuvant Therapy
Drug: Carboplatin — Given IV
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
Biological: Pegfilgrastim — Given IV
  Other Names: Filgrastim SD-01; GCSF-SD01; Neulasta

SUMMARY:
This phase I trial is studying the side effects of giving carboplatin and paclitaxel together with pegfilgrastim in treating patients with stage III or stage IV ovarian epithelial, fallopian tube, primary peritoneal, or carcinosarcoma cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving carboplatin and paclitaxel together with pegfilgrastim after surgery may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the feasibility of adjuvant dose-dense carboplatin and paclitaxel followed by pegfilgrastim, in terms of absence of grade 3 or 4 nonhematologic toxicities without major dose delays or additional hematological support (e.g., red blood cell or platelet transfusions or admission for febrile neutropenia), in patients with stage III-IV ovarian epithelial, fallopian tube, primary peritoneal cancer, or carcinosarcoma cancer.

SECONDARY OBJECTIVES:

I. Estimate the percentage of patients who develop ≥ grade 2 peripheral neurotoxicity from this regimen.

II. Estimate the clinical response rate in patients with measurable disease treated with this regimen.

III. Assess the toxicity of this regimen.

OUTLINE: This is a multicenter study.

Patients receive carboplatin IV and paclitaxel IV over 3 hours on day 1. Patients also receive pegfilgrastim subcutaneously on day 2. Treatment repeats every 2 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Primary peritoneal carcinoma
  * Fallopian tube carcinoma
  * Ovarian epithelial carcinoma
  * Carcinosarcoma
* Stage III or IV disease
* Previously untreated disease, except for mandatory prior surgery
* No ovarian epithelial carcinoma of low malignant potential (i.e., borderline carcinomas)
* GOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* No peripheral neuropathy (sensory or motor) ≥ grade 2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancies within the past 5 years except nonmelanoma skin cancer
* No septicemia, severe infection, or acute hepatitis
* No prior radiotherapy or chemotherapy
* No prior cancer treatment that would contraindicate study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-06; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who have greater than or equal to 1 dose-limiting toxicity, assessed by Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 12 weeks

SECONDARY OUTCOMES:
Number of patients with > grade 1 peripheral neuropathy based on the GOG neurotoxicity scale | Up to 1 year
Frequency and duration of objective response (complete and partial response) assessed by Response Evaluation Criteria for Solid Tumors (RECIST) | Up to 1 year
Grade of toxicity as assessed by CTCAE v3.0 | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, Principal Investigator — Gynecologic Oncology Group
Locations (11):
- United States (11):
  - University of California Medical Center At Irvine-Orange Campus, Orange, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington